CLINICAL TRIAL: NCT06296134
Title: Does Perineal Massage in Pregnancy Reduce the Levator Ani Muscle Co-activation?
Brief Title: Perineal Massage in Pregnancy to Reduce the Levator Ani Coactivation
Acronym: CO-LAM23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Universitaria Friuli Centrale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17501
Record Dates: First submitted 2024-02-14; First posted 2024-03-06 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Pelvic Floor Disorders; Levator Ani Syndrome
MeSH Terms: conditions — Pelvic Floor Disorders; Levator syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perineal massage (Experimental): participants randomized to this arm are asked to perform themselves the perineal massage once daily from 34 gestational weeks until delivery.
  Interventions: Behavioral: perineal massage
- standard care (No Intervention): participants randomized to this arm are asked to care for their pelvic floor according to the standard practice, which includes healthy diet, weight gain control, physical activity and voiding training therapy.

INTERVENTIONS:
Behavioral: perineal massage — women affected by LAM co-activation allocated to the intervention "perineal massage" are asked to perform the perineal massage once daily from 34 gestational weeks until delivery. Women are trained to correctly perform the perineal massage at 30 gestaitonal weeks.
  Arms: perineal massage

SUMMARY:
The goal of this clinical trial is to test the efficacy of the perineal massage in reducing the levator ani muscle (LAM) co-activation. This phenomenon is characterized by the LAM contraction rather than its relaxation during the Valsalva maneuver and it is associated with adverse obstetric outcome. Participants who co-activate will be enrolled and randomized in 2 groups: group A, where women themselves perform the perineal massage during the third trimester of pregnancy and group B, where women undergo the standard care. Researchers will compare these groups to see if the perineal massage is able to reduce LAM co-activation.

DETAILED DESCRIPTION:
The levator ani muscle has to relax instead of contracting during the pushing efforts in childbirth. However, some women consciously or unconsciously co-contract, or tighten, the levator ani muscle. This phenomenon is levator ani muscle co-activation. Recently, it has been shown that co-activation may be associated with unfavorable obstetric outcomes, such as prolonged second stages of labor and higher fetal head station in women with co-contraction.

Recently, a study assessing the correlation between levator ani muscle co-activation and perineal trauma has been published. This study found a significantly higher incidence of severe perineal trauma related to childbirth (i.e., third and fourth-degree lacerations and episiotomies) in women with levator ani muscle co-activation. This group of patients had approximately three times the risk of a vacuum-assisted vaginal delivery and five times the risk of developing a severe vagino-perineal laceration with potential involvement of the anal sphincter. Therefore, intervening in these patients with targeted measures to correct LAM co-activation in the third trimester of pregnancy might be promising.

Study design All women are informed about this study during the first trimester of pregnancy. During the anatomical scan, at 20-22 gestational weeks, women are screened for eligibility criteria, including: nulliparity, single pregnancy, fetus in cephalic presentation and fluency in Italian language. Women satisfying the inclusion criteria are asked to participate to this RCT. If women agree to participate in the study, an informed consent will be signed. Thereafter, a trans-perineal ultrasound will be performed in order to evaluate the presence of levator ani muscle co-activation. A medio-sagittal scan is obtained to identify the following landmarks: pubic symphysis, fetal head, rectum, and puborectal muscle. In this scan, the antero-posterior diameter of the anorectal angle (APD) is measured, which is the minimum distance between the postero-inferior border of the pubic symphysis and the anterior border of the puborectal muscle. This measurement is taken both at rest and during maternal pushing (Valsalva maneuver). Patients with co-activation will be identified by an APD during Valsalva that is smaller than the one observed at rest. Patients will be enrolled and randomized only in case of LAM co-activation.

A 1:1 randomization will be done using a specific function of Excel (preliminarily prepared by our Statistician). Women will be randomized in 2 arms: arm A is represented by the treatment "perineal massage", while arm B is represented by the "standard care".

At about 30 gestational weeks women randomized to arm A will be trained on how technically perform the perineal massage. Participants are instructed to do the perineal massage once daily from 34 gestational weeks until delivery, for at least 3 weeks continuously. By contrast, women randomized to arm B are informed on currently available recommendations to take care for pelvic floor in pregnancy. These recommendations include advices on healthy diet, physical activity and voiding training.

At 37-38 gestational weeks all randomized women are scanned again in order to measure the APD at rest and under Valsalva. All anthropometric and clinical data are collected and anonymized.

Intra-partum part of the study This part of the project involves data collection on labor, delivery, and neonatal outcomes. The labor and delivery care-providers operate blindly with respect to the antepartum ultrasound measurements.

The study was powered based on the primary endpoint, which is the 40% reduction in LAM co-activation at term after perineal massage therapy. It is necessary to randomize 58 subjects (29 women per group).

The primary outcome of this trial is to assess whether the intervention "perineal massage", compared to the standard care, is able to significantly reduce the levator ani co-activation. Secondary outcomes are the standardization of the perineal massage and the comparison of perineal trauma prevalence between the 2 arms.

ELIGIBILITY:
Inclusion Criteria: pregnant women with the following characteristics:

* nulliparous
* single pregnancy
* cephalic presentation of the fetus
* Italian language fluency

Exclusion Criteria:

* multiparous
* age < 18 y, age > 40 y
* previous urinary or fecal incontinence
* contraindications to vaginal delivery (such as placenta previa, vasa previa, etc)
* twin pregnancy
* language barrier
* BMI at or > 30

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the percentages of women without levator ani muscle co-activation after treatment or after standard care, evaluated at 37-38 weeks of gestation, using chi square test. | at 20 gestational weeks and at 37-40 gestational weeks
  All women who consent to participate in the study will be scanned through a trans-perineal ultrasound at 20 weeks. Co-activation is defined when the levator ani muscle antero-posterior diameter under Valsalva manueuver is lower than the same diameter measured at rest, with trans-perineal ultrasound.
  In case of LAM co-activation women will be recruited and randomized into two groups: the perineal massage group vs the standard care group. All randomized women will be evaluated with trans-perineal ultrasound for the levator ani muscle antero-posterior diameter measurement at 37-38 gestational weeks.
  To evaluate the effectiveness of the perineal massage, the percentages of women without LAM co-activation after treatment or after standard care, evaluated at 37-38 weeks, will be compared. For the comparison a chi square test will be used.

SECONDARY OUTCOMES:
Evaluation of significant differences in spontaneous or iatrogenic vaginal tears between the groups | immediately after fetus delivery
  The comparisons between groups will occur through chi-square tests for categorical variables and Student's t-tests for continuous variables.
  Vaginal tears are classified into first- degree, second- degree vaginal laceration, obstetric anal sphincter injury (OASI) and episiotomy
percentage of women who completely adhere to perineal massage, i.e. who perform the perineal massage once a day, at least 5 days a week, from 34 gestational weeks until delivery. | from 34 gestational weeks until the moment of delivery (between 37 weeks and 41 weeks and 3 days of gestation).
  for the effectiveness of perineal massage, participants in the "perineal massage" arm should perform the massage once a day, at least 5 days a week, from 34 gestational weeks until delivery. Participants will be asked to complete a diary, noting the days on which they perform the perineal massage.

CONTACTS AND LOCATIONS:
Locations (1):
- Serena Xodo, Udine, Italy

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: immediately after publication
Access Criteria: to gain access data requestors should contact the principal investigator: Serena Xodo, e-mail: serena.xodo@gmail.com

REFERENCES:
- [Background] Orno AK, Dietz HP. Levator co-activation is a significant confounder of pelvic organ descent on Valsalva maneuver. Ultrasound Obstet Gynecol. 2007 Sep;30(3):346-50. doi: 10.1002/uog.4082. PMID 17702054
- [Background] Kamel R, Montaguti E, Nicolaides KH, Soliman M, Dodaro MG, Negm S, Pilu G, Momtaz M, Youssef A. Contraction of the levator ani muscle during Valsalva maneuver (coactivation) is associated with a longer active second stage of labor in nulliparous women undergoing induction of labor. Am J Obstet Gynecol. 2019 Feb;220(2):189.e1-189.e8. doi: 10.1016/j.ajog.2018.10.013. Epub 2018 Oct 12. PMID 30321525
- [Background] Brunelli E, Del Prete B, Casadio P, Pilu G, Youssef A. The dynamic change of the anteroposterior diameter of the levator hiatus under Valsalva maneuver at term and labor outcome. Neurourol Urodyn. 2020 Nov;39(8):2353-2360. doi: 10.1002/nau.24494. Epub 2020 Aug 31. PMID 32865824
- [Background] Youssef A, Montaguti E, Dodaro MG, Kamel R, Rizzo N, Pilu G. Levator ani muscle coactivation at term is associated with longer second stage of labor in nulliparous women. Ultrasound Obstet Gynecol. 2019 May;53(5):686-692. doi: 10.1002/uog.20159. Epub 2019 Apr 2. PMID 30353589
- [Background] Youssef A, Brunelli E, Montaguti E, Di Donna G, Dodaro MG, Bianchini L, Pilu G. Transperineal ultrasound assessment of maternal pelvic floor at term and fetal head engagement. Ultrasound Obstet Gynecol. 2020 Dec;56(6):921-927. doi: 10.1002/uog.21982. PMID 31975450
- [Background] Youssef A, Brunelli E, Fiorentini M, Pilu G, El-Balat A. The correlation between levator ani co-activation and fetal head regression on maternal pushing at term. J Matern Fetal Neonatal Med. 2022 Dec;35(25):9654-9660. doi: 10.1080/14767058.2022.2050363. Epub 2022 Mar 13. PMID 35282757
- [Background] Beckmann MM, Stock OM. Antenatal perineal massage for reducing perineal trauma. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD005123. doi: 10.1002/14651858.CD005123.pub3. PMID 23633325